CLINICAL TRIAL: NCT05261958
Title: Effect of Speed, Agility and Quickness Training on Technical Skills in Football Players
Brief Title: Effect of Speed,Agility and Quickness Training on Technical Skills in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/01023/Sajjad Ali
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Physical Fitness
Keywords: Football, Technical skills, speed, agility, quickness

STUDY DESIGN:
Intervention Model Description: Two groups with randomization Assignment: High knee with mini hurdles, agility ring hops, 30 yard sprint, depth jumps, overhead ball drop
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): 1. Warm up and cool down (10 minutes before physical activity)
  2. Players will be given the SAQ training which includes
     * High Knees with Mini Hurdles.
     * 30 Yard Sprint.
     * Agility Ring Hops.
     * Ladder 2 in 2 out.
     * Depth Jumps.
     * Overhead Ball Drop Reaction Drill
  Interventions: Other: SAQ training
- Control Group (No Intervention): Players in this group did not undergo any interventional Programme rather than their daily routine work which includes:
  * Dumbbell squat
  * Dumbbell bicep arm curl
  * Burpee pull up
  * Medicine ball pushups
  * Sprints
  * HIIT on treadmill

INTERVENTIONS:
Other: SAQ training — interventions listed above were applied on the players which will improve running mechanics and impove speed power and agility in football players
  Other Names: High knee with mini hurdles; depth jumps; 30 yard sprint; Agility rings hops; Overhead ball drop
  Arms: Interventional Group

SUMMARY:
The study is designed to determine the effectiveness of Speed, Agility and Quickness training on technical skills in football players

DETAILED DESCRIPTION:
Football is a fast-paced, dynamic sport that requires expert movements. The goal of the game is to outscore your opponent in terms of goals scored. Players must perform a variety of expert movements, both with and without the ball, to achieve this goal. 'The learned ability to bring about predetermined results with utmost assurance, frequently with the least investment of time or energy or both,' according to an initial definition of talent. 'The constant output of goal-oriented movements, which are taught and unique to the job,' according to a more modern definition of competence. It is critical for players to have the fundamental motor abilities, such as running, agility, and acceleration, in order to learn and execute soccer skills effectively. Fundamental motor skills are seen as essential precursors or related factors to technical skills and therefore excellence in soccer.Furthermore, through a variety of soccer-specific activities, the SAQ training system consolidates speed, agility, and quickness. All exercises are carried out with appropriate biomechanical movement structures, resulting in significant energy and time savings. Aside from major abilities, power performance necessitates optimal joint mobility, dynamic balance, an appropriate locomotors system, and energy generation, among other things.

ELIGIBILITY:
Inclusion Criteria:

* Male players
* Age group of 18 years to 25 years.
* The study includes players, who are playing form 6 months to 1 year.

Exclusion Criteria:

* Players with any disability
* Injured players
* Players with psychological issues
* Players who are on any sort of medication

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male players of agr between 18years to 25 years and playing football from 6 months to 1 year
Enrollment: 50 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Shuttle Run test | 6 weeks
  Agility Shuttle Run is a test of agility, in which the participant runs back and forth between two parallel lines as fast as possible, picking up blocks of wood, for a total of 120 ft. A shuttle run time below four seconds is generally considered great, with the best players closer to the 3.8-second range, the total time is 4 seconds.
12 min run test | 6 weeks
  Place markers at set intervals around the track to aid in measuring the completed distance. Participants run for 12 minutes, and the total distance covered is recorded.
Speed | 6 weeks
  Set out a series of markers in a straight line at 0, 10, 20 and 30m. The player taking the test stands at the start, and the person timing stands on the 10m mark. On command, the player sprints through the 10m mark and the timer records the time they pass the marker. Repeat for 10m, and then do twice for 20m and 30m.
Vertical jump | 6 weeks
  The simplest method to measure an athlete's vertical jump is to get the athlete to reach up against a flat wall, with a flat surface under his/her feet and mark off the highest point he/she can reach flat-footed
Mcdonald Soccer skill test | 6 weeks
  A soccer ball is placed on a line, marked 9 feet from the wall. On the signal, "Go," the player kicks the ball against the wall as many times as possible in 30 seconds. The test score is the highest total of any three trials.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: No